CLINICAL TRIAL: NCT03825107
Title: Dichoptic Video Treatment for Amblyopia in Children Age 3-7 Years
Brief Title: Dichoptic Video Treatment for Amblyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Foundation of the Southwest (Other)
Responsible Party: Principal Investigator, Eileen Birch, Senior Research Scientist, Retina Foundation of the Southwest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dichoptic Video for Amblyopia
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Intervention Model Description: Parallel for primary outcome; crossover for longterm effectiveness
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patching (Active Comparator): 2 hours per day 7 days per week patching of the fellow eye
  Interventions: Other: patching
- Dichoptic Videos (Experimental): watching 6 dichoptic videos during each 2 week period
  Interventions: Other: Dichoptic videos

INTERVENTIONS:
Other: patching — covering the fellow eye with an eyepatch to force use of the amblyopic eye
  Other Names: occlusion therapy
  Arms: Patching
Other: Dichoptic videos — watching contrast-rebalanced dichoptic videos to allow the two eyes to work together
  Arms: Dichoptic Videos

SUMMARY:
1. To determine whether watching contrast-rebalanced dichoptic videos is effective in improving visual acuity and reducing interocular suppression in amblyopic children
2. To compare the amount of visual acuity improvement achieved with the videos to tha amount achieved with patching (standard treatment for amblyopia)

DETAILED DESCRIPTION:
Contrast-rebalanced binocular iPad tablet games (with fellow eye contrast reduced) have been shown to be an effective treatment for amblyopia. However, the games can be challenging for some of the youngest children and boring for some of the older children with amblyopia. To provide additional treatment options using the same contrast-rebalancing approach, we have processed animated videos to allow dichoptic viewing, with full contrast for the amblyopic eye and reduced contrast for the fellow eye. Children will be randomly assigned to watch dichoptic videos (experimental treatment) or patch 2 hours/day every day(standard-of-care amblyopia treatment) for 2 weeks. At the 2-week primary outcome visit, children in the patching group will cross over to the videos and return for a secondary outcome visit at 4 weeks. Families will have the option to continue with the vdeos for up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 3 to 7 years old
* Amblyopic eye visual acuity 20/32-20/125
* Fellow eye visual acuity 20/16-25
* Interocular visual acuity difference of at least 2 lines
* Anisometropia or corrected strabsimus (<5pd)
* in glasses at least 8 weeks or no change in visual acuity over two visits
* no prior binocular treatment
* must be able to see full video screen

Exclusion Criteria:

* prematurity of 8 weeks or more
* coexisting ocular or systemic disease
* developmental delay
* poor ocular alignment (>=5 pd)

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity of the amblyopic eye | Baseline vs 2 weeks
  HOTV (preferred) or picture chart

SECONDARY OUTCOMES:
Change in visual acuity of the amblyopic eye | Baseline vs 4 weeks, 6 weeks, and 8 weeks
  HOTV (preferred) or picture charts
Change in Stereoacuity | Baseline vs 2, 4, 6, 8 weeks
  Randot Preschool Stereoacuity test
Change in Contrast Balance Index | Baseline vs 2, 4, 6, 8 weeks
  Dichoptic Letter chart

CONTACTS AND LOCATIONS:
Overall Officials: Eileen E Birch, PhD, Principal Investigator — Retina Foundation of the Southwest
Locations (1):
- Eileen E Birch, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jost RM, Kelly KR, Birch EE. Risk of recurrence after cessation of dichoptic, binocular treatment of amblyopia. J AAPOS. 2023 Oct;27(5):298-300. doi: 10.1016/j.jaapos.2023.06.009. Epub 2023 Aug 23. PMID 37619861
- [Derived] Jost RM, Hudgins LA, Dao LM, Stager DR Jr, Luu B, Beauchamp CL, Hunter JS, Giridhar P, Wang YZ, Birch EE. Randomized clinical trial of streaming dichoptic movies versus patching for treatment of amblyopia in children aged 3 to 7 years. Sci Rep. 2022 Mar 9;12(1):4157. doi: 10.1038/s41598-022-08010-9. PMID 35264692

DOCUMENTS (2):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT03825107/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT03825107/SAP_001.pdf